CLINICAL TRIAL: NCT04815720
Title: A Phase 1b/2 Study of the Combination of Pepinemab and Pembrolizumab in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Pepinemab in Combination With Pembrolizumab in Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Acronym: KEYNOTE-B84
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vaccinex Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX15/2503-12; KEYNOTE-B84 (Other: Merck and Co., Inc.); MK3475-B84 (Other: Merck and Co., Inc.); VX15/2503 (Other: Vaccinex)
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck (HNSCC)
Keywords: Metastatic; Squamous Cell; Carcinoma; Recurrent; Pepinemab; Pembrolizumab; Head; Neck; VX15/2503; Solid Tumors; Immunotherapy; Progression-Free Survival (PFS); Objective Response Rate (ORR); Duration of Response (DOR); Pharmacokinetics (PK); Pharmacodynamics (PD); Immunogenicity; Biomarkers; Overall Survival (OS); Extent of Disease (EOD); Exploratory; Biopsy; T-Cell; Myeloid Suppressor Cells; ECG; KEYTRUDA®; MK3475-B84
MeSH Terms: conditions — Recurrence; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Carcinoma | interventions — pepinemab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This study will be conducted in 2 parts: a Safety Run-in phase and a Dose Expansion phase.
  The Safety Run-in phase will be based on the starting dose of 20 mg/kg pepinemab and a fixed dose of pembrolizumab (200 mg Q3W); 3 to 6 subjects will be treated at this pepinemab dose level. If the initial 20-mg/kg dose of pepinemab in combination with pembrolizumab is determined not to be well tolerated, the dose of pepinemab will be reduced to 15 mg/kg for an additional 3 subjects and a maximum of 6 subjects and then, potentially, to 10 mg/kg for a third group of 3 subjects and a maximum of 6 subjects.
  Once the recommended Dose Expansion phase dose is determined, a maximum of approximately 62 subjects will be treated with that dose of pepinemab combined with pembrolizumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- pepinemab + pembrolizumab (Experimental): Pepinemab will be administered at 20 mg/kg (with possible dose modifications to 15 mg/kg or 10 mg/kg, if the initial 20 mg/kg dose of pepinemab is determined not to be well tolerated) in combination with a fixed dose of 200 mg pembrolizumab, administered in separate IV infusions, Q3W.
  Interventions: Drug: pepinemab + pembrolizumab

INTERVENTIONS:
Drug: pepinemab + pembrolizumab — The Safety Run-in phase will begin at 20 mg/kg pepinemab with a fixed dose of 200 mg pembrolizumab. The dose of pepinemab may be reduced to 15 mg/kg or 10 mg/kg with a fixed dose of 200 mg pembrolizumab if the initial pepinemab dose of 20 mg/kg is found to not be well tolerated. Once a recommended phase II dose of pepinemab is determined it will be utilized in the Dose Expansion phase in combination with 200 mg pembrolizumab.
  Other Names: KEYTRUDA®

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of pepinemab in combination with pembrolizumab as first-line treatment and determine a recommended Phase 2 dose (RP2D) in patients with recurrent or metastatic head and neck squamous cell carcinoma (R/M HNSCC).

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the safety and tolerability of pepinemab in combination with pembrolizumab as first-line treatment and determine a recommended Phase 2 dose (RP2D) in patients with recurrent or metastatic head and neck squamous cell carcinoma (R/M HNSCC). The study will consist of a safety run in phase and a dose expansion phase.

The primary objective of the Safety Run-in phase of the study is to evaluate the safety and tolerability of pepinemab in combination with pembrolizumab as first-line treatment and determine a recommended Phase 2 dose (RP2D) for the dose-expansion phase enrolling subjects in patients with recurrent or metastatic head and neck squamous cell carcinoma (R/M HNSCC).

The primary objective of the Dose Expansion phase of the study is to evaluate objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 of the combination of pepinemab/pembrolizumab in immunotherapy naïve patients with R/M HNSCC.

The secondary objectives of the study are to evaluate progression-free survival (PFS) by RECIST 1.1 of the combination of pepinemab/pembrolizumab in immunotherapy naïve patients with R/M HNSCC, to evaluate the overall survival (OS), and to evaluate the duration of response (DOR).

The exploratory objectives of the study are to evaluate PFS, ORR, and DOR via the iRECIST criteria, to evaluate the pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of the combination, to investigate the relationship between treatment with pepinemab and pembrolizumab and certain biomarkers and the genomic signatures of baseline or archival tumor samples.

The Safety Run-in phase will enroll a minimum of 3 subject and a maximum of 18 subjects who will be treated with intravenous pepinemab IV (starting at 20 mg/kg, with potential dose modifications to 15 mg/kg or 10 mg/kg) and pembrolizumab at 200 mg IV, Q3W. The Dose Expansion phase of the study will enroll a maximum of approximately 62 subjects who will be treated with intravenous pepinemab administered IV at the RP2D, plus pembrolizumab 200 mg IV, Q3W.

Subjects will undergo evaluation for extent of disease (EOD) at baseline, week 9, every 6 weeks through year 1, and every 9 weeks thereafter. Subjects who discontinue study treatment will continue to be followed for survival every 12 weeks after safety follow-up (for up to approximately 2 years).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be ≥18 years of age.
2. Subjects or their legal representative must be able to provide written informed consent to participate in the trial prior to the performance of any study-specific procedures.
3. Subjects must have histologically or cytologically confirmed HNSCC; eligible histologies include SCC of the oropharynx, oral cavity, hypopharynx, and larynx.
4. Subjects must have PD-L1 IHC (including CPS score using an FDA approved test) testing completed within 6 months of screening or at screening.
5. Have measurable disease per RECIST 1.1 as assessed by the central imaging vendor or the local site investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Subjects must have locally advanced, recurrent or metastatic neoplastic disease that is not curable by currently available local therapies.
7. Subjects must have an Eastern Cooperative Oncology Group (ECOG) PS of 0 or1.
8. Subjects must have a life expectancy of at least 12 weeks.
9. Subjects must have adequate hematologic reserve based on the following:

   1. ANC ≥1,500/μL
   2. Platelet count >100,000/μL
   3. Hemoglobin >9 g/dL
10. Subjects must have adequate hepatic function based on the following:

    1. Total bilirubin <1.5 × upper limit of normal (ULN)
    2. Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤2.5 x ULN (≤5 x ULN for subjects with known hepatic metastases).
11. Subjects must have adequate renal function based on the following:

    1. Serum creatinine ≤1.5 × ULN; or
    2. Calculated creatinine clearance of >30 mL/min.
12. Human immunodeficiency virus (HIV) infected subjects must be on antiretroviral therapy (ART) and have a well-controlled HIV infection/disease defined as:

    1. Subjects on ART must have a CD4+ T cell count 350 cells/mm3 at time of screening
    2. Subjects on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 copies/mL or the lower limit of qualification (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks prior to screening
    3. Subjects on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks prior to study entry (Day 1).
13. Subjects with oropharyngeal cancer must have archival tissue available for p16 testing or be willing to undergo pre-study biopsy to obtain tissue for p16 testing.
14. All subjects must have archival or recently obtained tissue available for biomarker analysis.
15. Female subjects of childbearing potential must have a negative pregnancy test within 72 hours of first dose of study treatment. Female subjects of childbearing potential must use a highly effective mode of contraception or abstain from heterosexual activity for the duration of the trial and for 120 days following the last dose of study medication. A female is NOT of childbearing potential if she has undergone bilateral salpingoophorectomy or is menopausal, defined as an absence of menses for 12 consecutive months. Male subjects must agree to use highly effective contraception.

Exclusion Criteria:

1. Subjects with SCC of the nasopharynx.
2. Subjects who have received systemic treatment for recurrent or metastatic HNSCC; however, subjects who have received adjuvant systemic therapy or systemic therapy for locally advanced disease which was completed more than 6 months prior to study enrollment are eligible.
3. Subjects must have recovered from the effects of any prior radiation therapy or surgery.
4. Subjects who have received investigational therapy within 5 half-lives of the investigational agent or 4 weeks, whichever is shorter.
5. Subjects with primary immunodeficiency.
6. Subjects who require immunosuppressive therapy including, but not limited to, treatment with corticosteroids in pharmacologic doses (equivalent to ≥10 mg prednisone daily), cyclosporine, mycophenolate, azathioprine, methotrexate, adalimumab, infliximab, vedolizumab, tofacitinib, dupilumab, rituximab, etc.
7. Subjects with autoimmune conditions requiring treatment in the previous 2 years; however, subjects on replacement hormonal therapy alone for autoimmune endocrinopathies are eligible for enrollment.
8. Subjects with active central nervous system (CNS) metastases; however, subjects who have undergone radiation and/or surgery for the treatment of CNS metastases, who are neurologically stable and who are no longer taking pharmacologic doses of corticosteroids are eligible; subjects with leptomeningeal metastases are not eligible.
9. Has received prior radiotherapy within 2 weeks of start of study treatment. Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
10. Subjects with a prior malignancy (other than the malignancy under study) in the 2 years prior to enrollment; however, subjects with curatively treated nonmelanoma skin cancers, intra-epithelial cervical neoplasia or in situ carcinoma of the breast are eligible for enrollment.
11. Subjects with prior allogenic transplants.
12. Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis.
13. Subjects with an active infection requiring treatment with systemic antibiotics.
14. Subjects who are pregnant or lactating.
15. Subjects who have received treatment with a prior anti-PD-1 or anti-PD-L1, anti-CTLA-4, or anti-LAG3 agent or who have received prior treatment with pepinemab.
16. HIV-infected subjects with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
17. Subjects who are hepatitis B surface antigen positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to enrollment.

    Note: Subjects should remain on antiviral therapy throughout study intervention and follow local guidelines for HBV antiviral therapy post completion of study intervention.

    Hepatitis B screening tests are not required unless:
    1. Known history of HBV infection
    2. As mandated by local health authority.
18. Subjects with a history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening. Note: Subjects must have completed curative antiviral therapy at least 4 weeks prior to enrollment.

    Hepatitis C screening tests are not required unless:
    1. Known history of HCV infection
    2. As mandated by local health authority.
19. Subjects who have received a live vaccine within 30 days of study enrollment.
20. Current alcohol or drug abuse.
21. Subjects with any intercurrent medical condition where the known risks of participation in the trial outweigh any potential benefits; subjects with psychiatric or social circumstances that preclude responsible participation in the trial; subjects with severe nutritional deficiencies or marked hypoalbuminemia.
22. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
23. Inability to comply with visit schedule or other protocol requirements.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Treatment Emergent Adverse Events (TEAE's). | 2 Years
  TEAE's are defined as Adverse Events (AEs) with onset after date-time of first dose, or medical conditions present prior to the start of IMP but increased in severity or relationship after date-time of first dose of IMP.
Evaluation of RP2D | 2 Years
  Review number of subjects with incidence of laboratory abnormalities based on hematology, clinical chemistry, and urinalysis test results with consideration to ECG, vital sign measurements and physical examinations.
Efficacy Endpoint | 2 Years
  To be determined by the ORR of the combination pepinemab and pembrolizumab first-line treatment in patients with R/M HNSCC. This is defined as complete response (CR) or PR according to RECIST 1.1 from the first dose until documented confirmed disease progression.

SECONDARY OUTCOMES:
Duration of Response (DoR) | 2 Years
  To be measured from the first date of response (CR or PR) until the development of progressive neoplastic disease or death from any cause.
Overall Survival (OS) | 2 Years
  To be measured from the date of the first dose (Day 1 of Cycle 1) until death from any cause.
Progression Free Survival (PFS) | 2 Years
  To will be measured based on the RECIST 1.1 criteria from the date of enrollment until the development of progressive neoplastic disease or death from any cause.
Extent of Disease (EOD) | 2 Years
  To based on radiographic findings on computed tomography (CT) or magnetic resonance imaging (MRI) scan.
Pharmacokinetic (PK) Endpoints | 2 Years
  Area under the plasma concentration-time curve (AUC) from time zero to infinity (AUC0-∞).
Pharmacokinetic (PK) Endpoints | 2 Years
  AUC from time zero to the time of the last quantifiable concentration (AUC0-tlast).
Pharmacokinetic (PK) Endpoints | 2 Years
  Maximum observed plasma concentration (Cmax).
Pharmacokinetic (PK) Endpoints | 2 Years
  Time of the maximum observed plasma concentration (tmax).
Pharmacokinetic (PK) Endpoints | 2 Years
  Apparent plasma terminal elimination half-life (t1/2).
Pharmacokinetic (PK) Endpoints | 2 Years
  Apparent total plasma clearance (CL/F).
Pharmacokinetic (PK) Endpoints | 2 Years
  Apparent volume of distribution (Vz/F).
Immunogenicity Endpoint | 2 Years
  The incidence and severity of specific antidrug antibodies (ADA) to pepinemab.
Pharmacodynamic (PD) Endpoint | 2 Years
  Include receptor occupancy, cellular SEMA4D levels, and total soluble SEMA4D levels.

OTHER OUTCOMES:
On-Treatment Tumor Biopsies | 2 Years
  To be collected from the subjects who have readily accessible tumor tissue for determinations of T cell subpopulations and presence of MDSC and other myeloid suppressors (eg, M2 macrophage). These will be compared to pre-baseline tumor samples.
Serum and CSF Levels of Neuroinflammatory Cytokines | 2 Years
  IL-1, IL-2, IL-4, IL-5, IL-6, IL-10, IL-12, IL13,IFNγ, TNF-α, TGFβ
T- and B-Cell Quantitation by Flow Cytometry (TBNK) | 2 Years
  B cells, total count; Natural killer (NK) cells, total count; T cells, total count; Absolute CD4/CD8 count with ratio.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Highlands Oncology Group, PA - North Hills, Springdale, Arkansas
  - California Cancer Associates for Research and Excellence (CCARE)-Fresno, Fresno, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - AdventHealth Celebration, Celebration, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Siteman Cancer Center - Washington University Medical Campus, St Louis, Missouri
  - Northwell Health - Centers for Advanced Medicine, Lake Success, New York
  - University of Rochester, Rochester, New York
  - Messino Cancer Centers, Asheville, North Carolina
  - Gabrail Cancer Research Center, Canton, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Virginia Cancer Specialists - Fairfax, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher TL, Reilly CA, Winter LA, Pandina T, Jonason A, Scrivens M, Balch L, Bussler H, Torno S, Seils J, Mueller L, Huang H, Klimatcheva E, Howell A, Kirk R, Evans E, Paris M, Leonard JE, Smith ES, Zauderer M. Generation and preclinical characterization of an antibody specific for SEMA4D. MAbs. 2016;8(1):150-62. doi: 10.1080/19420862.2015.1102813. Epub 2015 Oct 2. PMID 26431358
- [Background] Dunn GP, Old LJ, Schreiber RD. The immunobiology of cancer immunosurveillance and immunoediting. Immunity. 2004 Aug;21(2):137-48. doi: 10.1016/j.immuni.2004.07.017. PMID 15308095
- [Background] Ribas A. Adaptive Immune Resistance: How Cancer Protects from Immune Attack. Cancer Discov. 2015 Sep;5(9):915-9. doi: 10.1158/2159-8290.CD-15-0563. Epub 2015 Aug 13. PMID 26272491
- [Background] Tumeh PC, Harview CL, Yearley JH, Shintaku IP, Taylor EJ, Robert L, Chmielowski B, Spasic M, Henry G, Ciobanu V, West AN, Carmona M, Kivork C, Seja E, Cherry G, Gutierrez AJ, Grogan TR, Mateus C, Tomasic G, Glaspy JA, Emerson RO, Robins H, Pierce RH, Elashoff DA, Robert C, Ribas A. PD-1 blockade induces responses by inhibiting adaptive immune resistance. Nature. 2014 Nov 27;515(7528):568-71. doi: 10.1038/nature13954. PMID 25428505
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Cowey CL, Lao CD, Schadendorf D, Dummer R, Smylie M, Rutkowski P, Ferrucci PF, Hill A, Wagstaff J, Carlino MS, Haanen JB, Maio M, Marquez-Rodas I, McArthur GA, Ascierto PA, Long GV, Callahan MK, Postow MA, Grossmann K, Sznol M, Dreno B, Bastholt L, Yang A, Rollin LM, Horak C, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Jul 2;373(1):23-34. doi: 10.1056/NEJMoa1504030. Epub 2015 May 31. PMID 26027431
- [Background] Clavijo PE, Moore EC, Chen J, Davis RJ, Friedman J, Kim Y, Van Waes C, Chen Z, Allen CT. Resistance to CTLA-4 checkpoint inhibition reversed through selective elimination of granulocytic myeloid cells. Oncotarget. 2017 Jun 11;8(34):55804-55820. doi: 10.18632/oncotarget.18437. eCollection 2017 Aug 22. PMID 28915554
- [Background] Janssen BJ, Robinson RA, Perez-Branguli F, Bell CH, Mitchell KJ, Siebold C, Jones EY. Structural basis of semaphorin-plexin signalling. Nature. 2010 Oct 28;467(7319):1118-22. doi: 10.1038/nature09468. Epub 2010 Sep 26. PMID 20877282
- [Background] Tamagnone L, Artigiani S, Chen H, He Z, Ming GI, Song H, Chedotal A, Winberg ML, Goodman CS, Poo M, Tessier-Lavigne M, Comoglio PM. Plexins are a large family of receptors for transmembrane, secreted, and GPI-anchored semaphorins in vertebrates. Cell. 1999 Oct 1;99(1):71-80. doi: 10.1016/s0092-8674(00)80063-x. PMID 10520995
- [Background] Ch'ng ES, Kumanogoh A. Roles of Sema4D and Plexin-B1 in tumor progression. Mol Cancer. 2010 Sep 21;9:251. doi: 10.1186/1476-4598-9-251. PMID 20858260
- [Background] Younis RH, Han KL, Webb TJ. Human Head and Neck Squamous Cell Carcinoma-Associated Semaphorin 4D Induces Expansion of Myeloid-Derived Suppressor Cells. J Immunol. 2016 Feb 1;196(3):1419-29. doi: 10.4049/jimmunol.1501293. Epub 2016 Jan 6. PMID 26740106
- [Background] Chen Y, Zhang L, Lv R, Zhang WQ. Overexpression of Semaphorin4D indicates poor prognosis and prompts monocyte differentiation toward M2 macrophages in epithelial ovarian cancer. Asian Pac J Cancer Prev. 2013;14(10):5883-90. doi: 10.7314/apjcp.2013.14.10.5883. PMID 24289594
- [Background] Ch'ng E, Tomita Y, Zhang B, He J, Hoshida Y, Qiu Y, Morii E, Nakamichi I, Hamada K, Ueda T, Aozasa K. Prognostic significance of CD100 expression in soft tissue sarcoma. Cancer. 2007 Jul 1;110(1):164-72. doi: 10.1002/cncr.22764. PMID 17520683
- [Background] Clavijo PE, Friedman J, Robbins Y, Moore EC, Smith E, Zauderer M, Evans EE, Allen CT. Semaphorin4D Inhibition Improves Response to Immune-Checkpoint Blockade via Attenuation of MDSC Recruitment and Function. Cancer Immunol Res. 2019 Feb;7(2):282-291. doi: 10.1158/2326-6066.CIR-18-0156. Epub 2018 Dec 4. PMID 30514791
- [Background] Evans EE, Jonason AS Jr, Bussler H, Torno S, Veeraraghavan J, Reilly C, Doherty MA, Seils J, Winter LA, Mallow C, Kirk R, Howell A, Giralico S, Scrivens M, Klimatcheva K, Fisher TL, Bowers WJ, Paris M, Smith ES, Zauderer M. Antibody Blockade of Semaphorin 4D Promotes Immune Infiltration into Tumor and Enhances Response to Other Immunomodulatory Therapies. Cancer Immunol Res. 2015 Jun;3(6):689-701. doi: 10.1158/2326-6066.CIR-14-0171. Epub 2015 Jan 22. PMID 25614511
- [Background] Leonard JE, Fisher TL, Winter LA, Cornelius CA, Reilly C, Smith ES, Zauderer M. Nonclinical Safety Evaluation of VX15/2503, a Humanized IgG4 Anti-SEMA4D Antibody. Mol Cancer Ther. 2015 Apr;14(4):964-72. doi: 10.1158/1535-7163.MCT-14-0924. Epub 2015 Feb 5. PMID 25657333
- [Background] LaGanke C, Samkoff L, Edwards K, Jung Henson L, Repovic P, Lynch S, Stone L, Mattson D, Galluzzi A, Fisher TL, Reilly C, Winter LA, Leonard JE, Zauderer M. Safety/tolerability of the anti-semaphorin 4D Antibody VX15/2503 in a randomized phase 1 trial. Neurol Neuroimmunol Neuroinflamm. 2017 Jun 16;4(4):e367. doi: 10.1212/NXI.0000000000000367. eCollection 2017 Jul. PMID 28642891
- [Background] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428
- [Background] Dudley ME, Wunderlich JR, Yang JC, Sherry RM, Topalian SL, Restifo NP, Royal RE, Kammula U, White DE, Mavroukakis SA, Rogers LJ, Gracia GJ, Jones SA, Mangiameli DP, Pelletier MM, Gea-Banacloche J, Robinson MR, Berman DM, Filie AC, Abati A, Rosenberg SA. Adoptive cell transfer therapy following non-myeloablative but lymphodepleting chemotherapy for the treatment of patients with refractory metastatic melanoma. J Clin Oncol. 2005 Apr 1;23(10):2346-57. doi: 10.1200/JCO.2005.00.240. PMID 15800326
- [Background] Hunder NN, Wallen H, Cao J, Hendricks DW, Reilly JZ, Rodmyre R, Jungbluth A, Gnjatic S, Thompson JA, Yee C. Treatment of metastatic melanoma with autologous CD4+ T cells against NY-ESO-1. N Engl J Med. 2008 Jun 19;358(25):2698-703. doi: 10.1056/NEJMoa0800251. PMID 18565862
- [Background] Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol. 2005;23:515-48. doi: 10.1146/annurev.immunol.23.021704.115611. PMID 15771580
- [Background] Okazaki T, Maeda A, Nishimura H, Kurosaki T, Honjo T. PD-1 immunoreceptor inhibits B cell receptor-mediated signaling by recruiting src homology 2-domain-containing tyrosine phosphatase 2 to phosphotyrosine. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):13866-71. doi: 10.1073/pnas.231486598. Epub 2001 Nov 6. PMID 11698646
- [Background] Zhang X, Schwartz JC, Guo X, Bhatia S, Cao E, Lorenz M, Cammer M, Chen L, Zhang ZY, Edidin MA, Nathenson SG, Almo SC. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity. 2004 Mar;20(3):337-47. doi: 10.1016/s1074-7613(04)00051-2. PMID 15030777
- [Background] Chemnitz JM, Parry RV, Nichols KE, June CH, Riley JL. SHP-1 and SHP-2 associate with immunoreceptor tyrosine-based switch motif of programmed death 1 upon primary human T cell stimulation, but only receptor ligation prevents T cell activation. J Immunol. 2004 Jul 15;173(2):945-54. doi: 10.4049/jimmunol.173.2.945. PMID 15240681
- [Background] Sheppard KA, Fitz LJ, Lee JM, Benander C, George JA, Wooters J, Qiu Y, Jussif JM, Carter LL, Wood CR, Chaudhary D. PD-1 inhibits T-cell receptor induced phosphorylation of the ZAP70/CD3zeta signalosome and downstream signaling to PKCtheta. FEBS Lett. 2004 Sep 10;574(1-3):37-41. doi: 10.1016/j.febslet.2004.07.083. PMID 15358536
- [Background] Riley JL. PD-1 signaling in primary T cells. Immunol Rev. 2009 May;229(1):114-25. doi: 10.1111/j.1600-065X.2009.00767.x. PMID 19426218
- [Background] Parry RV, Chemnitz JM, Frauwirth KA, Lanfranco AR, Braunstein I, Kobayashi SV, Linsley PS, Thompson CB, Riley JL. CTLA-4 and PD-1 receptors inhibit T-cell activation by distinct mechanisms. Mol Cell Biol. 2005 Nov;25(21):9543-53. doi: 10.1128/MCB.25.21.9543-9553.2005. PMID 16227604
- [Background] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Background] Hirano F, Kaneko K, Tamura H, Dong H, Wang S, Ichikawa M, Rietz C, Flies DB, Lau JS, Zhu G, Tamada K, Chen L. Blockade of B7-H1 and PD-1 by monoclonal antibodies potentiates cancer therapeutic immunity. Cancer Res. 2005 Feb 1;65(3):1089-96. PMID 15705911
- [Background] Blank C, Brown I, Peterson AC, Spiotto M, Iwai Y, Honjo T, Gajewski TF. PD-L1/B7H-1 inhibits the effector phase of tumor rejection by T cell receptor (TCR) transgenic CD8+ T cells. Cancer Res. 2004 Feb 1;64(3):1140-5. doi: 10.1158/0008-5472.can-03-3259. PMID 14871849
- [Background] Weber J. Immune checkpoint proteins: a new therapeutic paradigm for cancer--preclinical background: CTLA-4 and PD-1 blockade. Semin Oncol. 2010 Oct;37(5):430-9. doi: 10.1053/j.seminoncol.2010.09.005. PMID 21074057
- [Background] Strome SE, Dong H, Tamura H, Voss SG, Flies DB, Tamada K, Salomao D, Cheville J, Hirano F, Lin W, Kasperbauer JL, Ballman KV, Chen L. B7-H1 blockade augments adoptive T-cell immunotherapy for squamous cell carcinoma. Cancer Res. 2003 Oct 1;63(19):6501-5. PMID 14559843
- [Background] Spranger S, Koblish HK, Horton B, Scherle PA, Newton R, Gajewski TF. Mechanism of tumor rejection with doublets of CTLA-4, PD-1/PD-L1, or IDO blockade involves restored IL-2 production and proliferation of CD8(+) T cells directly within the tumor microenvironment. J Immunother Cancer. 2014 Feb 18;2:3. doi: 10.1186/2051-1426-2-3. eCollection 2014. PMID 24829760
- [Background] Curran MA, Montalvo W, Yagita H, Allison JP. PD-1 and CTLA-4 combination blockade expands infiltrating T cells and reduces regulatory T and myeloid cells within B16 melanoma tumors. Proc Natl Acad Sci U S A. 2010 Mar 2;107(9):4275-80. doi: 10.1073/pnas.0915174107. Epub 2010 Feb 16. PMID 20160101
- [Background] Pilon-Thomas S, Mackay A, Vohra N, Mule JJ. Blockade of programmed death ligand 1 enhances the therapeutic efficacy of combination immunotherapy against melanoma. J Immunol. 2010 Apr 1;184(7):3442-9. doi: 10.4049/jimmunol.0904114. Epub 2010 Mar 1. PMID 20194714
- [Background] Nomi T, Sho M, Akahori T, Hamada K, Kubo A, Kanehiro H, Nakamura S, Enomoto K, Yagita H, Azuma M, Nakajima Y. Clinical significance and therapeutic potential of the programmed death-1 ligand/programmed death-1 pathway in human pancreatic cancer. Clin Cancer Res. 2007 Apr 1;13(7):2151-7. doi: 10.1158/1078-0432.CCR-06-2746. PMID 17404099
- [Background] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- See also: 19. Keytruda® (pembrolizumab) prescribing information (June 2020; injection for intravenous use). — https://www.merck.com/product/usa/pi_circulars/k/keytruda/keytruda_pi.pdf.